CLINICAL TRIAL: NCT06039553
Title: A Comprehensive Research of Pediatric Heart Failure -- A Self-control Study of Pulmonary Artery Banding for the Improvement of Left Ventricular Function in Pediatric Heart Failure
Brief Title: Study of Pulmonary Artery Banding for the Improvement of Left Ventricular Function in Pediatric Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Peking University First Hospital (Other); Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Shoujun Li, Director of Congenital Heart Surgery Center, China National Center for Cardiovascular Diseases
Other Study IDs: 2022-1-4032-2
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure Congenital
Keywords: congenital heart disease; pulmonary artery banding
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Artery Banding Group: Patient in this group will undergo pulmonary artery banding surgery for congenital heart disease.
  Interventions: Procedure: pulmonary artery banding

INTERVENTIONS:
Procedure: pulmonary artery banding — Patient in this group will undergo pulmonary artery banding surgery for congenital heart disease.

SUMMARY:
The goal of this observational study is to learn about the safety and effectiveness of pulmonary artery banding(PAB) therapy in pediatric heart failure(PHF) patients.

The main questions it aims to answer are:

* Can PAB therapy improve left ventricular(LV) function in PHF patients especially refractory PHF.
* Can the complications caused by the PAB therapy be clinically acceptable? Participants underwent PAB therapy will be required to underwent echocardiography, electrocardiograms, complete blood counts, biochemical tests, and measurements of N-terminal pro-brain natriuretic peptide (NT-proBNP) follow-up before the initiation of PAB and at 1 month, 3 months, and 6 months after PAB surgery. Researchers will compare the LV function 6 months after PAB suergey and the preoperative ones to see if there is improvement.

ELIGIBILITY:
Inclusion Criteria:

* patients younger than 14 years of age
* congenital heart failure (LVEF<55%, or LVFS<25%)

Exclusion Criteria:

* single ventricle
* congenital heart disease without anatomical correction
* Patients with heart failure requiring ventricular assist or cardiac synchronization therapy
* Patients with severe pulmonary hypertension (pulmonary arterial pressure >6 Wood·U)
* Patients with severe liver and kidney failure
* Patients who are allergic to related medications
* Patients with symptomatic hypotension who cannot tolerate related drugs
* Refuse to sign the informed consent or refuse to participate in this experiment

Max Age: 14 Years | Sex: All
Age Groups: Child
Study Population: paitent younger than 14 years of age with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of heart failure | after 6 months of PAB surgery
  During follow-up visits, echocardiographic examination is conducted to measure the left ventricular function. If LVEF falls under 55%, it is recorded as a recurrence.

SECONDARY OUTCOMES:
NT-proBNP level | after 6 months of PAB surgery
  The trend in NT-proBNP levels.
Incidence rate of drug adverse reactions | after 6 months of PAB surgery
  The incidence of abnormalities in complete blood count, electrolytes, liver and kidney function, and cardiac enzymes.
Readmission rate for heart failure | after 6 months of PAB surgery
  During follow-up visits, readmission for heart failure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shoujun Li, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No